CLINICAL TRIAL: NCT02938702
Title: Active Surveillance on Papillary Thyroid Microcarcinoma
Status: Active, not recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Young Joo Park, Professor, Seoul National University Hospital
Other Study IDs: 2520160010
Record Dates: First submitted 2016-02-17; First posted 2016-10-19 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Thyroid Cancer; Papillary Thyroid Microcarcinoma
Keywords: Active surveillance
MeSH Terms: conditions — Thyroid Neoplasms; Papillary Thyroid Microcarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Active surveillance: Group with active surveillance of their PTC
- Surgery: Group who underwent surgery after diagnosis of PTC

SUMMARY:
The study is a multi-center prospective cohort study of active surveillance in papillary thyroid cancer with low risk. The purpose of the study is to observe natural course of low risk papillary thyroid cancer in Korean population, and comparison of prognosis between active surveillance group and conventional surgery group. Patient will be well informed about their choice of active surveillance or surgery.

ELIGIBILITY:
Inclusion Criteria:

* who agreed to the agreement form
* who is older than 18 years old
* who was diagnosed by fine needle aspiration or needle biopsy of Bethesda category V or VI
* whose thyroid cancer is smaller than 1 cm length

Exclusion Criteria:

* who cannot routinely follow-up according to the study schedule
* who was diagnosed by fine needle aspiration or needle biopsy of Bethesda category I, II, III, or IV.
* who have hyperthyroidism which needs treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient aged older than 18 years with papillary thyroid microcarcinoma less than 1 cm in length, who did not meet the exclusion criteria from Seoul National University Hospital, National Cancer Center, Seoul National University Bundang Hospital, and Borame Medical Center.
Sampling Method: Probability Sample
Enrollment: 1211 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Rate of Progression of Thyroid Papillary Microcarcinoma | 5 years
  rate of progression: tumor size increase of ≥3 mm in at least one dimension, tumor size increase of ≥2 mm in at least two dimensions, suspected organ involvement during the follow-up, such as trachea, esophagus, nerves, vessels, or muscles in imaging study including high-resolution ultrasonography, or pathological diagnosis of lymph node/distant metastasis

SECONDARY OUTCOMES:
Comparison of Progression Rate between Active Surveillance and Surgery Group | 5 years
  Which group had higher progression rate; progression defined as whether tumor size increases more than 3 mm in diameter, or tumor involves new lymph nodes, or metastasis occurs

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee JY, Kim JH, Kim YK, Lee CY, Lee EK, Moon JH, Choi HS, Yul H, Cho SW, Kim SJ, Lee KE, Park DJ, Park YJ. US Predictors of Papillary Thyroid Microcarcinoma Progression at Active Surveillance. Radiology. 2023 Oct;309(1):e230006. doi: 10.1148/radiol.230006. PMID 37906009
- [Derived] Hwang H, Choi JY, Yu HW, Moon JH, Kim JH, Lee EK, Kim YK, Lee CY, Cho SW, Chung EJ, Ryu CH, Ryu J, Yi KH, Park DJ, Lee KE, Park YJ, Kim SJ, Jung YS. Surgical Outcomes in Patients With Low-risk Papillary Thyroid Microcarcinoma From MAeSTro Study: Immediate Operation Versus Delayed Operation After Active SurveillanceA Multicenter Prospective Cohort Study. Ann Surg. 2023 Nov 1;278(5):e1087-e1095. doi: 10.1097/SLA.0000000000005841. Epub 2023 Mar 13. PMID 36912439
- [Derived] Lee EK, Moon JH, Hwangbo Y, Ryu CH, Cho SW, Choi JY, Chung EJ, Jeong WJ, Jung YS, Ryu J, Kim SJ, Kim MJ, Kim YK, Lee CY, Lee JY, Yu HW, Hah JH, Lee KE, Lee YJ, Park SK, Park DJ, Kim JH, Park YJ. Progression of Low-Risk Papillary Thyroid Microcarcinoma During Active Surveillance: Interim Analysis of a Multicenter Prospective Cohort Study of Active Surveillance on Papillary Thyroid Microcarcinoma in Korea. Thyroid. 2022 Nov;32(11):1328-1336. doi: 10.1089/thy.2021.0614. PMID 36205563
- [Derived] Hwangbo Y, Choi JY, Lee EK, Ryu CH, Cho SW, Chung EJ, Hah JH, Jeong WJ, Park SK, Jung YS, Kim JH, Kim MJ, Kim SJ, Kim YK, Lee CY, Lee JY, Lee YJ, Yu HW, Park DJ, Ryu J, Park YJ, Lee KE, Moon JH. A Cross-Sectional Survey of Patient Treatment Choice in a Multicenter Prospective Cohort Study on Active Surveillance of Papillary Thyroid Microcarcinoma (MAeSTro). Thyroid. 2022 Jul;32(7):772-780. doi: 10.1089/thy.2021.0619. PMID 35698288
- [Derived] Moon JH, Ryu CH, Cho SW, Choi JY, Chung EJ, Hah JH, Hwangbo Y, Jeong WJ, Jung YS, Kim JH, Kim MJ, Kim SJ, Kim YK, Lee CY, Lee EK, Lee JY, Lee KE, Lee YJ, Lee Y, Yu HW, Park DJ, Ryu J, Park YJ. Effect of Initial Treatment Choice on 2-year Quality of Life in Patients with Low-risk Papillary Thyroid Microcarcinoma. J Clin Endocrinol Metab. 2021 Mar 8;106(3):724-735. doi: 10.1210/clinem/dgaa889. PMID 33248442